CLINICAL TRIAL: NCT06729892
Title: Feasibility of Closed-loop TCI Based on New BIS Baseline in the Presence of Low Dose of Esketamine: a Randomized Controlled Equivalence Trial.
Brief Title: Feasibility of Closed-loop TCI Based on New EEG Baseline in the Presence of Low Dose of Esketamine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: bo xu (Other)
Responsible Party: Sponsor-Investigator, bo xu, Doctor; Chief director., Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GuangzhouGH; 62076253 (Other Grant/Funding Number: Bo Xu); 82472110 (Other Grant/Funding Number: Bo Xu)
Record Dates: First submitted 2024-12-07; First posted 2024-12-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: General Anesthesia With Propofol; Closed-Loop
Keywords: eskemine; close-loop TCI; EEG; depth of anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adjusted-group (Experimental): After administering esketamine at low dose , this group adjusted drug dosage under closed-loop control based on the new BIS baseline(50＋N).
  Interventions: Drug: Esketamine at low dose; Device: new BIS baseline
- Non-adjusted group (Experimental): After administering esketamine at low dose, this group adjusted drug dosage under closed-loop control based on the original BIS baseline(50).
  Interventions: Drug: Esketamine at low dose; Device: original BIS baseline
- control group (Placebo Comparator): This group adjusted drug dosage under closed-loop control based on the original BIS baseline(50) with an equivalent volume of saline.
  Interventions: Drug: an equivalent dose of saline; Device: original BIS baseline

INTERVENTIONS:
Drug: Esketamine at low dose — Esketamine at low dose was administered(0.2mg· kg-1, 5 ug· kg-1 continuous infusion) and drug dosage was adjusted(propofol and remifentanil) based on the new BIS baseline ( calculated from the pilot study).
  Arms: Adjusted-group; Non-adjusted group
Device: new BIS baseline — Close-loop TCI control was under new BIS baseline(calculated from pilot study) in the presence of esketamine at low dose.
  Arms: Adjusted-group
Drug: an equivalent dose of saline — An equivalent dose of saline was given and closed-loop control stared.
  Arms: control group
Device: original BIS baseline — Drug dosage was adjused under close-loop control based on original BIS baseline.
  Arms: Non-adjusted group; control group

SUMMARY:
The propofol-remifentanil closed-loop TCI system based on EEG guidance has been clinically verified, which enables more precise anesthetic dosing. As an adjunct to anesthesia, esketamine has been shown to stabilize hemodynamics, reduce opioid use, and reduce postoperative nausea and vomiting. However, due to its specific electroencephalographic excitatory effect, esketmine's clinical use in close-loop system has been limited. The aim of this experiment was to determine the specific impact of esketamine on EEG and thus obtain a new EEG baseline for close-loop system, which can broaden the application of close-loop TCI system in combination with other drugs.

DETAILED DESCRIPTION:
The trial is devided into two phases. In the first phase, we statistically analyzed and calculated the changes of BIS by collecting a sample size of EEG changes after administering low dose of esketamine. We used 0.2 mg/kg as a loading dose and followed by a rate of 5ug/kg/min as esketamine administration and observe the changes in BIS each for 30 minutes.

In the second phase, we obtain the BIS quantification value N with the addition of a small dose of esketamine in the first phase and thus obtain a new EEG baseline 50+N. By comparing this EEG-adjusted group with the control group, which run the close-loop system based on original BIS baseline without esketamine, whether the closed-loop system can be better applied based on the new BIS baseline under low dose of esketamine.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18~27kg· m-2;
* American Society of Anesthesiologists (ASA)physical status I~II;
* Undergoing elective laparoscopic surgery.

Exclusion Criteria:

* Known or suspected neurological diseases, tumors, stroke, degenerative neurological diseases, epileptic seizures, serious head injuries, cognitive disorders, post-traumatic stress disorder, mental illnesses, severe depression, psychosis, etc.;
* Contraindications to ketamine, propofol or remifentanil;
* Use of psychotropic drugs within the past 7 days;
* History of drug abuse or drug addiction within the past 30 days or during pregnancy;
* Current participation in any other studies involving other drugs or devices.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
BIS, % of time within ± 10 units of the BIS setpoint during closed-loop control | time of closed-loop control, started from 10 min after esketamine administration and lasted for 50 min
  % of time within ± 10 units of the BIS setpoint is the most commonly used metric to evaluate performance of closed-loop control.

SECONDARY OUTCOMES:
drug consumption | time of closed-loop control, started from 10 min after esketamine administration and lasted for 50 min
  drug consumption of propofol and remifentanil
hemodynamic changes during closed-loop control | time of closed-loop control, started from 10 min after esketamine administration and lasted for 50 min
Postoperative recovery assessment | time to BIS>80, time to regain spontaneous breathing, time to answering questions and time to extubate
VAS | time from PACU administration to transfer out from PACU.
  visual analgesic score, one of a most commonly used critieria of pain intensity. VAS ranges from 0~10, 0~3 indicates slight or no pain; 4~6 indicates Moderate pain; 7~10 indicates severe pain.
extra analgesic drugs usage | From transfer into and out PACU
occurrance of nausea and vomiting, shivering | From transfer into and out PACU
intraoperative awareness assessment, 15-item quality of recovery (QoR-15) | From postoperative day 1st to day 7th.
  Intraoperative awareness is assessed by modified Brice questionnaire; This questionnaire consists of 5 questions. Level of Intraoperative awareness ranges from 0~5. The QoR-15 questionnaire is composed of 15 questions, including physical comfort (5 items), emotional state (4 items), physical independence (2 items), psychological support (2 items), and pain(2 items). The higher of the QoR-15 scores, the better of the quality of recovery after surgery (range is 0 to 150 points).

CONTACTS AND LOCATIONS:
Overall Officials: BO xu, doctor, chief director, Study Director — department of anesthesiology, southern theater general hospital of PLA, Guangzhou, China.

IPD SHARING:
Plan to Share IPD: No